CLINICAL TRIAL: NCT00656773
Title: A Randomized, Double-blind Comparison of Morphine and Sufentanil for Treatment of Prehospital Traumatic Severe Acute Pain.
Brief Title: A Randomized, Double-blind Comparison of Morphine and Sufentanil for Prehospital Traumatic Severe Acute Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07 139 03; N° EUDRACT 2007-004049-14
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Acute Pain
Keywords: morphine, sufentanil, acute pain, opioid, Prehospital Emergency Care
MeSH Terms: conditions — Acute Pain | interventions — Sufentanil; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Sufentanil
- 2 (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Sufentanil — 0.15 μg/kg, IV following by 0.075 μg/kg every 3 minutes during 15 minutes
  Arms: 1
Drug: Morphine — 0.15 mg/kg, IV following by 0.075 mg/kg every 3 minutes during 15 minutes
  Arms: 2

SUMMARY:
Obtaining high-quality analgesia in prehospital patients with severe pain is an important treatment objective for medical team. Opioids are recognized as the treatment of choice for relief of severe acute pain. Recommended initial analgesia of patients with severe acute pain, defined as a visual analog scale or a numerical rating scale (NRS) score of 60/100 or higher, in a prehospital setting in France consists of the administration of opioids by the medical staff of mobile intensive care units. The intravenous administration of morphine is usually considered as the gold standard for postoperative acute pain relief because of its rapid transport from the blood to target tissues after intravenous injection, its long-lasting analgesic effect without any plateau, and its well-known pharmacokinetics. Nevertheless, the short-acting opioid sufentanil might be preferable to the traditional long-acting morphine for prehospital analgesia because of its even faster onset of action and shorter duration than morphine. There is no study, to our knowledge, comparing the clinical efficacy of sufentanil vs morphine in a prehospital setting. This randomized double-blind group clinical trial is designed to determine the best intravenous opioid titration protocol by comparing sufentanil and morphine for medical prehospital treatment of adult patients with severe acute pain. Eligible patients with a numerical rating scale (NRS) score of 60/100 or higher will be randomly allocated to receive either 0.15 µg/kg sufentanil then 0.075 µg/kg every 3 minutes (group A) or 0.15 mg/kg morphine then 0.075 mg/kg every 3 minutes (group B) intravenously. The decision to provide opioid analgesia including titration of subsequent doses of narcotic is the responsibility of physicians and intravenous analgesia will be given and titrated according to the pain score every 3 minutes. The drugs will be administered by the physician from syringes of similar appearance prepared by the nurse who is not otherwise involved in the study. The protocol-defined primary outcome measure is the percentage of patients with pain relief (with a NRS score of 30/100 or lower) 15 minutes after the first injection. Secondary outcomes include pain score comparisons every 3 minutes within the first 30 minutes and comparison of adverse events. The physician blinded to the analgesic treatment groups will do all assessments of patients. The safety evaluation will include non invasive monitoring of blood pressure, heart rate, respiratory rate, oxygen saturation by pulse oximetry (Spo2), and a sedation scale (0, patient is awake; 1, patient is with intermittent sleeping; 2, patient is sleeping, awakened by verbal stimulation; 3, patient is sleeping, awakened by tactile stimulation; 4, patient is not aroused by stimulation) at these periods. Fifteen minutes after the first injection, overall patient and investigator satisfaction with analgesia was recorded.

DETAILED DESCRIPTION:
Obtaining high-quality analgesia in prehospital patients with severe pain is an important treatment objective for medical team. Opioids are recognized as the treatment of choice for relief of severe acute pain. Recommended initial analgesia of patients with severe acute pain, defined as a visual analog scale or a numerical rating scale (NRS) score of 60/100 or higher, in a prehospital setting in France consists of the administration of opioids by the medical staff of mobile intensive care units. The intravenous administration of morphine is usually considered as the gold standard for postoperative acute pain relief because of its rapid transport from the blood to target tissues after intravenous injection, its long-lasting analgesic effect without any plateau, and its well-known pharmacokinetics. Nevertheless, the short-acting opioid sufentanil might be preferable to the traditional long-acting morphine for prehospital analgesia because of its even faster onset of action and shorter duration than morphine. There is no study, to our knowledge, comparing the clinical efficacy of sufentanil vs morphine in a prehospital setting. This randomized, controlled, double-blind, parallel group clinical trial is then designed to determine the best intravenous opioid titration protocol by comparing sufentanil and morphine for medical prehospital treatment of adult patients with severe acute pain. Eligible patients with a numerical rating scale (NRS) score of 60/100 or higher will be randomly allocated to receive either 0.15 µg/kg sufentanil then 0.075 µg/kg every 3 minutes (group A) or 0.15 mg/kg morphine then 0.075 mg/kg every 3 minutes (group B) intravenously. The decision to provide opioid analgesia including titration of subsequent doses of narcotic is the responsibility of physicians and intravenous analgesia will be given and titrated according to the pain score every 3 minutes. The drugs will be administered by the physician from syringes of similar appearance prepared by the nurse who is not otherwise involved in the study. The protocol-defined primary outcome measure is the percentage of patients with pain relief (with a NRS score of 30/100 or lower) 15 minutes after the first injection. Secondary outcomes include pain score comparisons every 3 minutes within the first 30 minutes and comparison of adverse events. The physician blinded to the analgesic treatment groups will do all assessments of patients. The safety evaluation will include non invasive monitoring of blood pressure, heart rate, respiratory rate, oxygen saturation by pulse oximetry (Spo2), and a sedation scale (0, patient is awake; 1, patient is with intermittent sleeping; 2, patient is sleeping, awakened by verbal stimulation; 3, patient is sleeping, awakened by tactile stimulation; 4, patient is not aroused by stimulation) at these periods. Fifteen minutes after the first injection, overall patient and investigator satisfaction with analgesia (pain relief classified as excellent, good, mild, or weak) was recorded. We will analyze the primary and secondary end points using the intention-to-treat method.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* with a severe traumatic acute pain defined by an NRS score of 60/100 or higher at randomization.

Exclusion Criteria:

* Patient-reported history of chronic respiratory, renal, or hepatic insufficiency
* known opioid or acetaminophen allergies
* treatment of chronic pain or treatment with opioids
* incapacity to understand the NRS
* hypotension (defined as a systolic blood pressure b90 mm Hg,bradypnea of less than 12/min, oxygen desaturation of less than 90%, seizures or a Glasgow Coma Scale score of less than 14
* pregnancy
* drug addiction
* Patients who had already received an analgesic, including aspirin or acetaminophen within 6 hours (either by self-administration or by another physician in attendance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The protocol-defined primary outcome measure is the percentage of patients with pain relief (with a NRS score of 30/100 or lower) 15 minutes after the first injection. | 15 minutes after the first injection.

SECONDARY OUTCOMES:
Secondary outcomes include pain score comparisons every 3 minutes within the first 30 minutes, comparison of adverse events and overall patient and investigator satisfaction with analgesia. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: DUCASSE Jean-louis, MD, Principal Investigator — UH Toulouse
Locations (1):
- U H Toulouse Samu 31, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bounes V, Barthelemy R, Diez O, Charpentier S, Montastruc JL, Ducasse JL. Sufentanil is not superior to morphine for the treatment of acute traumatic pain in an emergency setting: a randomized, double-blind, out-of-hospital trial. Ann Emerg Med. 2010 Nov;56(5):509-16. doi: 10.1016/j.annemergmed.2010.03.020. Epub 2010 Apr 10. PMID 20382445